CLINICAL TRIAL: NCT01621269
Title: A 12-month, Open-label, Multicenter Study to Evaluate the Efficacy and Safety of Fingolimod in the Treatment of Relapsing-remitting Multiple Sclerosis Patients With Neutralizing Antibodies to Interferon Beta
Brief Title: ENGYNE Exploring Gilenya in Patients With Neutralizing Antibodies Against Interferon
Acronym: ENGYNE
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CFTY720DDE12
Record Dates: First submitted 2012-04-24; First posted 2012-06-18 (Estimated); Last update posted 2017-04-20 (Actual); Status verified 2014-09

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; MS; Fingolimod; Gilenya; Neutralizing Antibodies; NAb
MeSH Terms: conditions — Multiple Sclerosis | interventions — Fingolimod Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Fingolimod (Experimental)
  Interventions: Drug: Fingolimod

INTERVENTIONS:
Drug: Fingolimod

SUMMARY:
Study to evaluate efficacy of fingolimod in patients with neutralizing antibodies over 12 months

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged 18-65 years
* Subjects with relapsing remitting MS defined by 2010 revised McDonald criteria
* Patients with Expanded Disability Status Scale (EDSS) score of 0-6.5
* Interferon-beta (IFN-β) treatment for at least 18 months.
* Positive IFN-NAb titer at screening or within 6 months prior to screening
* Patients with disease activity despite treatment with IFN-ß measured by gadolinium-enhancing lesions on T1-weighted images on MRI using a triple-dose gadolinium protocol and/or new or newly enlarging T2 lesions (T2 lesions: compared to a reference MRI performed within the last 18 months)

Exclusion Criteria:

* patients with previous or current disease of immune system
* active infections
* cardiovascular risk patients
* Patients unable to undergo MRI scans, including claustrophobia or history of hypersensitivity to gadolinium-DTPA

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-06; Primary Completion 2014-06 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Number of patients with active MRI lesions | 12 months
  number of patients with neutralizing antibodies against IFN-ß with reduction of number of combined unique active lesions on brain MRI (CUAL) defined as those lesions that are new or recurrent or enlarging on T2-weighted scans or those that are new and taking Gd-enhancement on T1-weighted scans, avoiding double counting

SECONDARY OUTCOMES:
Number of patients with adverse events | 12 months
  safety of fingolimod as measured by number of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals